CLINICAL TRIAL: NCT01723020
Title: A Phase 1 First-in-Human Study Evaluating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 232 in Adult Subjects With Advanced Solid Tumors or Multiple Myeloma
Brief Title: A Phase 1 Study Evaluating AMG 232 in Advanced Solid Tumors or Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20120106
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Advanced Malignancy; Advanced Solid Tumors; Cancer; Oncology; Oncology Patients; Tumors; Glioblastoma; Multiple Myeloma
Keywords: Solid Tumors; Multiple Myeloma
MeSH Terms: conditions — Neoplasms; Glioblastoma; Multiple Myeloma | interventions — 2-(5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-(1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AMG 232 (Experimental): AMG 232 is an anti-cancer agent.
  Interventions: Drug: AMG 232

INTERVENTIONS:
Drug: AMG 232 — Given an an oral tablet in escalating doses.

SUMMARY:
First in human, open-label, sequential dose escalation and expansion study of AMG 232 in subjects with advanced solid tumors or multiple myeloma

DETAILED DESCRIPTION:
Study Design: This is an open-label, dose exploration study evaluating AMG 232 in subjects with advanced p53WT solid tumors or multiple myeloma. The study will be conducted in 2 parts: Part 1 - Dose Exploration (parts 1a, 1b and 1c) and Part 2 - Dose Expansion. Part 1a is aimed at evaluating the safety, tolerability, PK and PD of AMG 232 and determining the MTD of a 7-day once daily (QD) dosing schedule in subjects with advanced solid tumors using a practical continuous reassessment method (CRM). Part 1b will evaluate the safety and tolerability of 3-day QD dosing schedule (or alternate dosing schedule based upon emerging data) with a particular emphasis on evaluating the tolerability of daily doses equal to or higher than the part 1a MTD in subjects with solid tumors or multiple myeloma. Part 1c will evaluate the safety and tolerability of 7-day twice daily (BID) dosing schedule with daily cumulative doses equal to or higher than the part 1a MTD in subjects with solid tumors. The dose expansion part of the study (Part 2) can open once the MTD has been determined in Part 1a. Part 2, part 1b and part 1c can be explored in parallel. The dose expansion part will consist of up to 85 additional subjects with specific tumors harboring MDM2 amplification (liposarcoma [LPS], gliobastoma [ GBM ] and all other solid tumors) or potentially harboring MDM2 overexpression (ER+ metastatic breast cancer) and a group of subjects with multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years old
* Pathologically documented, definitively diagnosed, advanced solid tumor that is refractory to standard treatment, or which no standard therapy is available, or the subject refuses standard therapy or multiple myeloma
* Willing to undergo pre-dose core needle tumor biopsies or bone marrow aspirate for subjects with multiple myeloma.
* Ability to take oral medications and willing to record daily adherance to investigational product
* Adequate hematological, renal, hepatic, and coagulation laboratory assessments

Exclusion Criteria:

* Active brain metastases
* For solid tumor-History or presence of hematological malignancies unless curatively treated with no evidence of disease for greater than or equal to 5 years
* Active infection requiring intravenous (IV) antibiotics
* Anti-tumor therapy
* Therapeutic or palliative radiation therapy within 30 days of starting treatment
* Currently enrolled in another investigational device or drug study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-12-27 (Actual); Primary Completion 2017-03-15 (Actual); Study Completion 2017-09-25 (Actual)

PRIMARY OUTCOMES:
Safety of AMG 232 | 36 months
  Subject incidence of adverse events, dose limiting toxicities, and clinically significant changes in vital signs, weight, ECGs and clinical laboratory tests

SECONDARY OUTCOMES:
Objective Tumor Response | 36 months
  Duration of overall response and duration of stable disease measured by CT or MRI and assessed per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1, for multiple myeloma using IMWG response criteria

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (13):
- United States (8):
  - Research Site, Santa Monica, California
  - Research Site, Norwalk, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, Hackensack, New Jersey
  - Research Site, New Brunswick, New Jersey
  - Research Site, New York, New York
  - Greenville Hospital System, Greenville, South Carolina
  - Research Site, Greenville, South Carolina
- France (2):
  - Research Site, Lyon
  - Research Site, Villejuif
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Rotterdam
  - Research Site, Utrecht

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com